CLINICAL TRIAL: NCT03934281
Title: Study of the Value of Using a Honey Dressing Compared to the Use of a Standard Dressing on the Toe Amputation Wound in the Diabetic Patient
Acronym: MELIDIAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Metropole Savoie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHMS17001
Record Dates: First submitted 2019-04-04; First posted 2019-05-01 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Diabete Mellitus; Amputation; Amputation Wound; Toe (Toes); Wound
MeSH Terms: conditions — Diabetes Mellitus; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAS dressing (Active Comparator): Patients included in the "HAS dressing" arm will receive the best available dressing according to the HAS recommendations. HAS is the french National Authority for Health (HAS) .
  Interventions: Device: HAS recommendation dressing
- Honey dressing (Experimental): the honey used in this study is the Melectis G dressing. This is a combination of thyme honey (99.8%) and hyaluronic acid (0.2%).
  The patient will benefit from the honey dressing until complete healing and/or until the end of the study (maximum 12 months).
  Interventions: Device: Honey dressing Melectis G

INTERVENTIONS:
Device: Honey dressing Melectis G — The protocol includes rinsing the wound with the saline, gently drying the edge of the wound, applying a thin Mélectis®G film to the entire wound surface and covering with a secondary dressing.
  Dressings will be rehabilitated based on the evolution of the wound and clinical judgement of the investigator or nurse at home as recommended.
  Arms: Honey dressing
Device: HAS recommendation dressing — Patients included in the standard arm will receive the best available dressing according to the HAS recommendations.
  Dressings will be rehabilitated based on the evolution of the wound and clinical judgement of the investigator or nurse at home as recommended.
  Arms: HAS dressing

SUMMARY:
Numerous scientific publications in France and internationally have described the healing, anti-bacterial, anti-oxidant, anti-inflammatory and immuno-modulating properties of honey.

Honey is effective in the management of many infected or uninfected post-surgical wounds.

This study focuses on post surgical wounds after toe amputation in diabetic patients.

The main objective of this study is to compare the rate of epidermisation at six months for these wounds, between honey dressing and other dressing devices used according to the french Haute Autorité de Santé (HAS) recommendations

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients
* Patients who have had an amputation of one or more toes within four days prior to inclusion without having the second dressing rehabilitated
* Written informed consent.

Exclusion Criteria:

* Known hypersensitivity to honey, hyaluronic acid, guar gum, pectin and/or zinc oxide.
* Insipid Diabètes
* patient eligible for a dressing by Vacuum Assisted Closure therapy (VAC therapy)
* transmetatarsal amputation
* Patient with sutured wound
* Patient already included in the study, for a previous amputation for wich the wound has not healed.
* Failure to comply with protocol requirements
* Person protect by article L1121-5 to L1121-8 of the French Health Public.
* Patient include in an other clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
Epidermization rate at 6 months. | 6 months after amputation
  the relative difference between the volume of the wound in mm3 during the first rehabilitation of the post-operative dressing (J0) and this volume six months after (M6), on the volume of the wound in mm3 at J0. (TM6 = (VD0 - VM6) /VD0)

SECONDARY OUTCOMES:
Epidermization rate at 12 months | 12 months after amputation
  the relative difference between the volume of the wound in mm3 during the first rehabilitation of the post-operative dressing (J0) and this volume 12 months after (M12), on the volume of the wound in mm3 at J0. (T = (VD0 - VM12) /VD0)
pain during dressing change: verbal scale of pain | inclusion, 1month, 2 months, 3months, 4months, 5 months, 6 months,7months,8months, 8months ,9months 10months, 11months, 12 months after amputation up to cicatrization
  verbal scale of pain. this scale measures the pain of patient. the ranges are 0 to 4.
average length of wound cicatrization | from date of amputation until the date of the first documented complete cicatrization, assessed up to 12 months
  The average length of wound healing in case of complete healing before the end of the study.
the satisfaction of professionals for the use of honey dressing | 12 months after amputation or at study completion, whichever came first
  the level of satisfaction of all professionals involved in the rehabilitation of the honey dressing, will be evaluated with a Likert scale.The Likert scale, which falls under our definition of a survey scale, is a 5 point scale that ranges from one extreme attitude to another, like "extremely likely" to "not at all likely." They include a moderate or neutral midpoint.
Epidermization rate at 1 month | 1 month after amputation
  the relative difference between the volume of the wound in mm3 during the first rehabilitation of the post-operative dressing (J0) and this volume 1 month after (M1), on the volume of the wound in mm3 at J0. (T = (VD0 - VM1) /VD0)
Epidermization rate at 2 months | 1 month after amputation
  the relative difference between the volume of the wound in mm3 during the first rehabilitation of the post-operative dressing (J0) and this volume 2 months after (M2), on the volume of the wound in mm3 at J0. (T = (VD0 - VM2) /VD0)

CONTACTS AND LOCATIONS:
Locations (1):
- Hélène Blaise, Chambéry, France

IPD SHARING:
Plan to Share IPD: No